Weaning From Mechanical Ventilation in Neurological Patients

NCT03128086

Date: March 3, 2017

INTRODUCTION

A high percentage of patients with acute neurological disease require invasive

mechanical ventilation (MV) to isolate the airway, to provide adequate oxygenation and to

prevent aspiration of gastric content (1-3). During weaning from MV, a spontaneous breathing

trial (SBT) is realized before extubation in order to assess patient's capacity to breath (4-6),

and reducing the risk of extubation failure. The extubation failure is associated with a

prolonged length of stay in the intensive care unit (ICU) and in the hospital, as well as, more

risk of infections and higher mortality (7). In neurological patients, a successful SBT can not

predict exactly the success of extubation (8-10). It is necessary both the assessment of muscle

strength and the ability to keep the airway clearance capacity to ensure success of extubation

(8-15).

The results obtained with the application of weaning protocols in neurological patients

are not conclusive (16), with the exception of one clinical trial (17). A meta-analysis concluded

that the establishment of weaning protocols in subjects in a medical-surgical unit reduced the

duration of MV by 25%, weaning time by 78% and ICU stay by 10%. These results support the

use of weaning protocols in patients undergoing MV (18).

In this study we try to demonstrate that the use of a protocol-directed weaning in

neurological patients will reduce the rate of extubation failure and associated complications.

The primary objective is to reduce the failure rate of extubation. As secondary objectives we

are going to analyse the incidence of infections, need for tracheostomy, duration of MV, length

of ICU and hospital stay, and mortality at ICU, hospital and 90 days.

MATERIAL AND METHODS

A prospective interventionist no randomized study will be conducted in a medical-

surgical ICU. Patients 18 years or older with acute medical or surgical neurological disease

[acute ischaemic or haemorrhagic stroke, acute subarachnoid haemorrhage, traumatic brain

trauma, metabolic encephalopathy (toxic, infectious as encephalitis or meningitis), scheduled

neurosurgical surgery with a prolonged MV, and status epileptics], will be included. Exclusion

Criteria: scheduled neurosurgical surgery (duration of MV <24 hours), neuromuscular disease,

1

spinal cord injury, tracheostomized, inability to be evaluated, severe multiple traumatic injuries evaluated by the Injury Severity Score (19), direct extubation and self-extubation, patients who died during their ICU stay (without a trail of weaning), and patients transferred to another hospital.

At ICU admission, the following variables will be collected: age, sex, body mass index, comorbidities, prognosis severity scale by Simplified Acute Physiological Score (SAPS) 3, Organ failure by Sequential Organ Failure Assessment (SOFA) (at ICU admission and 5 days after admission), reason for MV, the level of consciousness by Glasgow Coma Scale (GCS) at the time of intubation and where it was performed. During the ICU stay, all neurological treatments and procedures such as treatment of intracranial hypertension (manitol or hypertonic saline, hyperventilation, decompressed craniotomy), cranial tomography (CT) scanner, external ventricular drainage, intracranial pressure sensor, cerebral arteriography, will be collected. The infectious complications (ventilator-associated pneumonia, tracheobronchitis, urinary tract infection, bacteraemia,) will be registered during the ICU stay.

To be included into study, subject undergoing mechanical ventilation will meet the following conditions: no or minimal sedation (propofol $\leq 1$ mg/kg/h o midazolam $\leq 0.1$ mg/kg/h), with spontaneous ventilatory stimulus, absence of intracranial hypertension, Glasgow Coma Score (GCS)> 9 (motor> 4 points), noradrenaline  $\leq 0.2$ mcgr/kg/min, (fraction of inspired oxygen)FiO2  $\leq 0.5$  (positive end-expiratory pressure) PEEP of 5cmH20, no intervention scheduled in the next 48 hours, maximal inspiratory pressure (MIP)< -20cmH20 (20), occlusion pressure (P0.1) >6mmHg with support pressure of 7cmH20 and 0 cmH20 of positive end-expiratory pressure (Z-PEEP).

**Protocol study (study group)**. The subject will be connected to MV in a pressure support ventilation (PSV) mode, which will be gradually reduced (until a level de pressure support of 10 cmH20 above 5 cmH20 of PEEP). After, the subject will be disconnected from the ventilator and a SBT will begin through the connexion of the subject to a T-tube and a source of oxygen (21). Haemodynamic parameters [systolic blood pressure (SBP), heart rate (HR)], and respiratory parameters [respiratory rate (RR), partial pressure of carbon dioxide (paCO2), partial pressure of oxygen to fraction of inspired oxygen ratio (paO2/FiO2), and pH through blood gas analysis and saturation of oxyhemoglobin (SaO2) by pulse oximetry], and neurological parameters (means by GCS) will be collected during final period of pressure support ventilation (before disconnection) and at onset (5 minutes) and final (between 30 to 120 minutes) of SBT (22). A once daily SBT will be established in all the subjects until they

were extubated. A failure SBT will be considered with more than 2 criteria: pa02<50-60mmHg with FiO2  $\leq$  0.5 (or SaO2 <90%), paCO2 > 50 mmHg, pH <7.35, RR > 35bpm, HR > 140 bpm, SBP > 180mmHg, cardiac arrhythmias during SBT, dyspnea, and increased use of accessory muscles (6). If the SBT fails, the subject will reconnect to MV. A successful SBT is defined as absence of whatever of variables above defined. *Airway clearance capacity*. Otherwise, if the SBT is successful, the ability to maintain airway will be analysed by the following variables: Number of aspirations of secretions/8-h nursing shift (No pass-0, 1 pass-1, 2 passes-2,  $\geq$  3 passes-3), cough capacity (strong -0, mild-1, weak-2, absent-3), appearance of secretions [viscosity (liquid-0, frothy-1, thick-2, dry-3) and colour of secretions (clear-0, brown- 1, yellow-2, green-3), and finally, the presence of gag reflex (strong- 0, moderate- 1, weak- 2, absent- 3). A score  $\leq$ 8 was considered as adequate to keep the permeability of airway (4). Then the subject will be extubated and connected to venturi mask with FiO2 of 0.4. In case of extubation failure, the patient will be reintubated. The use of non-invasive ventilation is not considered in this study (neither prevention of extubation failure nor in case of extubation failure).

Conventional weaning (control group). Subjects in the control group will receive weaning from MV according to the usual procedure, by reducing level of PSV. Then a SBT will be performed through a T-tube (the same parameters as protocol study will be collected) and subsequent extubation of the patient if there is a successful SBT. The criteria for SBT and for extubation failure are the same than in the study group. In case of extubation failure, non-invasive ventilation will be not considered, but it left to the discretion of the attending physician.

STATISTIC ANALYSIS. Based upon previous results (10), the authors considered that the need for an intubation could be reduced by 13% (6) [26% in the control group vs. 13% in the study group]. The estimated sample size was 109 patients in each group (confidence interval  $[1-\alpha]$  = 95% (P=0.05) and power  $[1-\beta]$  = 80%). A comparative analysis was conducted by using the Student's t-test or the Mann-Whitney test for a comparison of the quantitative variables for the parametric and non-parametric characteristics, respectively. For the qualitative variables, we used the Chi-Square statistic or Fisher's exact test. A statistical significance was reached if P<0.05. The cumulative probability of survival was compared by using a Kaplan-Meier estimation of survival and a Log-Rank Test to compare both of the groups. Intention-to-treat

analysis will be realized. The data will be analysed with the aid of the statistical package SPSS 22.0.

## REFERENCE

- Esteban A, Anzueto A, Frutos F, Alía I, Brochard L, Stewart ThE, Benito S, Epstein SK, Apezteguía C, Nightingale P, Arroliga AC, Tobin MJ, for the Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation. JAMA 2002; 287-355
- 2. Pelosi P, Ferguson ND, Frutos-Vivar F, Anzueto A, Putensen Ch, Raymondos K, et al for the Ventila Study Group. Management and outcome of mechanically ventilated neurologic patiens. Crit Care Med 2011; 39: 1482-1492
- 3. Guerrero López F, Fernández-Mondéjar E. Extubación de pacientes neurocríticos con bajo nivel de conciencia. Un problema a resolver. Med Intensiva 2000; 24: 304-306
- 4. Coplin WM, Pierson DJ, Cooley KD, Newell DW, Rubenfeld GD. Implications of extubation delay in brain-injured patients meeting standar weaning criteria. Am J Respir Crit Care Med 2000; 161:1530-1536
- 5. MacIntyre N, Cook D, Ely EW Jr, Epstein SK, Fink JB, Hubmayr RD, et al. Evidence-Based Guidelines for weaning and discontinuing ventilatory support: A collective task force facilitated by American College of Chest Physicians, The American Association ofr Respiratory Care, And the American College of Criticial Care Medicine. Respir Care 2002; 47:69-90.
- 6. Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, et al. Statement of the Sixth International Consensus Conference on Intensive Care Medicine. Weaning from mechanical ventilation. Eur Respi J 2007; 29:1033-1056
- 7. Epstein SK, Ciubotaru RL, Wong JB. Effect of failed extubation on the outcome of mechanical ventilation. Chest 1997; 112:186-192

- 8. King Ch, Moores LK, Epstein SK. Should patients be able to follow commands prior to extubation?. Respir Care 2009; 55:56-62
- 9. Vallverdú I, Calaf N, Subirana M, Net A, Benito S, Mancebo J. Clinical characteristics, respiratory functional parameters and outcome of a two hours T-piece trial in patients weaning from mechanical ventilation. Am J Respir Crit Care Med 1998; 158: 1855-1862
- 10. Belenguer-Muncharaz A, Mateu-Campos ML, Ferrándiz-Sellés MD, Vidal-Tegedor B, Altaba-Tena S, Casero-Roig P, Micó-Gómez ML, Álvaro-Sánchez R, Rodríguez-Martínez EA, De Léon-Belmar J. Análisis retrospectivo sobre la extubación en pacientes con patología neurológica aguda. Medicina Intensiva 2015; 32: 1
- 11. Ko R, Ramos L, Chalela JA. Conventional weaning parameters do not predict extubation failure in neurocritical care patients. Neurocrit Care 2009; 10: 269-273
- 12. Castro A, Cortopassi F, Sabbag R, Torre-Bouscoulet L, Kümpel C, Ferreira E. Evaluación de la musculatura respiratoria en la predicción del resultado de la extubación de pacientes con ictus. Arch Bronconeumol 2012; 48: 274-279
- 13. Khamiees M, Raju P, DeGirolamo A, Amoateng-Adjepong Y, Manthous C. Predictors of extubation outcome in patients who have successfully completed a spontaneous breathing trial. Chest 2001; 120: 1262-1270
- 14. Salam A, Tillckdharry L, Amoateng-Adjepong Y, Manthous CA. Neurologic status, cough, secretions and extubation outcomes. Intensive Care med 2004; 30:1334-1339
- 15. Beuret P, Roux C, Auclair A, Nourdine K, Kaaki M, Carton MJ. Interest of an objective evaluation of cough during weaning from mechanical ventilation. Intensive Care Med 2009; 35: 1090-1093
- 16. Namen AM, Ely EW, Tatter SB, Case D, Lucia MA, Smith A, et al. Predictors of successful extubation in neurosurgical patients. Am J Respir Crit Care Med 2001; 163:658-664
- 17. Navalesi P, Frigerio P, Moretti M, Sommariva M, Vesconi S, Baiardi P, et al. Rate of reintubation in mechanically ventilated neurosurgical and neurologic patients: Evaluation of a systematic approach to weaning and extubation. Crit Care Med 2008; 36: 2986-2992

- 18. Blackwood B, Alderdice F, Burns K, Cardwell Ch, Lavery G, O'Halloran. Use of weaning protocols for reducing duration of mechanical ventilation in critically ill adult patients:

  Cochrane systematic review and meta-analysis. BMJ 2011; 342:c7237 doi:10.1136/bmj.c/23/
- 19. Baker CC, Degutis LC. Injury Severity Score. Infect surgical 1986;5: 243-245
- 20. Caruso P, Friederich C, Denari S, Ruiz S, Deheinzelin D. The unidirectional valve is the best method to determine maximal inspiratory pressure during weaning. Chest 1999; 115:1096-1101
- 21. Esteban A, Alía I, Gordo F, Fernández R, Solsona JF, Vallverdú I, et al. Extubation outcome after spontaneous breathing trials with T-Tube or pressure support ventilation. Am J Respir Crit Care Med 1997; 156: 459-465
- 22. Esteban A, Alía I, Tobin MJ, Gil A, Gordo F, Vallberdú I, et al. Effects of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation.

  Am J Respir Crit Care Med 1999; 159: 512-518